CLINICAL TRIAL: NCT01366937
Title: Assessment of Vitamin B12 Bioavailability From Egg
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Lindsay H. Allen, ARS USDA WHNRC
Other Study IDs: 200715660-2
Record Dates: First submitted 2009-01-16; First posted 2011-06-06 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Bioavailability of Vitamin B12 From Chicken Eggs
Keywords: vitamin B12; egg; 14C; fecal excretion

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Plasma, serum, buffy coat, urine, stool
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of this study is that chicken eggs can be enriched in vivo with 14C-B12 and fed to healthy human subjects to determine B12 bioavailability from eggs.

The goal of this research is to enrich eggs in vivo with radioactively labeled vitamin B12 to a level that allows us to feed the enriched eggs to humans and determine how much of the vitamin B12 is digested and absorbed into the body. This will tell us if eggs are a good dietary source of vitamin B12. Importantly, sensitive technology available at the Lawrence Livermore National Laboratories allows us to measure very low amounts of radioactive vitamin B12. This allows us to do this experiment with a level of radioactive B12 that is not harmful to animals or humans. The results of the investigators first experiment indicate that the investigators can inject radioactively labeled vitamin B12 into a laying hen and detect the radioactive vitamin B12 in the eggs at a level sufficient for feeding to humans in a bioavailability study.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy subjects, adequate B12 status and absorptive capacity and the availability to complete the protocol.

Exclusion Criteria:

* any chronic health disorder, anemia of any kind, renal insufficiency, and pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults, 18 y or older
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Fecal enrichment of 14C | Over the course of 8 days after dosing with 14C labeled egg

CONTACTS AND LOCATIONS:
Overall Officials: Linday H Allen, PhD, Principal Investigator — ARS, USDA, WHNRC; Marjorie G Garrod, PhD, Study Chair — ARS, USDA, WHNRC
Locations (1):
- Usda, Ars, Whnrc, Davis, California, United States